CLINICAL TRIAL: NCT04634201
Title: Effect of Probiotics in Addition to Dental Brushing on Gum Inflammation and Oral Microbiota in Patients With Fixed Orthodontic Appliances
Brief Title: Effect of Probiotics on the Periodontal Status of Orthodontic Patients
Acronym: POP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Sunstar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019_14; 2020-A02179-30 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Periodontal Health; Gingivitis
Keywords: Gingivitis; oral microbiota; salivary biomarkers; probiotics
MeSH Terms: conditions — Gingivitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Dietary Supplement: Oral probiotics (L. reuteri)
- control group (Sham Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral probiotics (L. reuteri) — administration of probiotic containing tablets twice daily after tooth brushing for 3 months
  Arms: Experimental group
Dietary Supplement: Placebo — administration of a placebo twice daily after tooth brushing for 3 months
  Arms: control group

SUMMARY:
Gingival inflammation (gingivitis) is commonly reported in teenagers with fixed orthodontic devices (FOD). Indeed, FODs promote the accumulation of plaque and interfere with the efficacy of tooth brushing. According to in vitro and in vivo studies, the administration of oral probiotic bacteria including Lactobacillus reuteri may reduce the number of periodontal pathogens in saliva and dental plaque. A recent systematic review shows a positive effect of probiotics in addition to tooth brushing in the treatment of periodontitis. However, there is insufficient data regarding the effect of probiotics in the prevention of gum diseases. The aim of this double-blind randomized placebo-controlled study is to assess the effect of probiotics, in addition to dental brushing, on gum inflammation and the composition of the oral microbiota in teenagers with fixed orthodontic appliances

ELIGIBILITY:
Inclusion Criteria:

* adolescents aged 12 to 16 benefiting from social security coverage
* in good general health in brushing and taking treatments
* Have FODs
* who consent to the study and whose parents have given their consent
* suitable for orthodontic treatment in view of his oral state

Exclusion Criteria:

* inability to obtain informed consent
* use of another probiotic or toothpaste / antiseptic mouthwash ≤ 1 month before inclusion
* allergy or hypersensibiliity to the active substance or to any of the excipients listed in the Gum® PerioBalance® user guide)
* no history of antibiotic therapy, antiseptic mouthwash ≤ 1 month before inclusion
* medical contraindication (immunosuppression, pathology requiring prophylactic antibiotic therapy before dental care)
* physiological, pathological condition, medication or behavior that may have repercussions on the oral cavity (eg: pregnancy, diabetes, antiepileptics, tobacco)
* oral state requiring other priority care (untreated cavities, untreated active periodontitis, progressive recession)

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Variation of gingival index (Löe Silness) between baseline and 6 months | At 6 months

SECONDARY OUTCOMES:
bleeding on probing (BOP) score (% of BOP sites) | At Baseline, at 3 months and 6 months
plaque index (O'leary) | At Baseline, at 3 months and 6 months
dysbiosis index | At Baseline, at 3 months and 6 months
  Shannon-weaver, alpha rarefaction, beta diversity
level of salivary markers of inflammation - | At Baseline, at 3 months and 6 months
compliance level record | At Baseline, at 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevimy AGOSSA, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Salengro - Chu Lille, Lille, France